CLINICAL TRIAL: NCT05515887
Title: Evaluation on the Influence of Shenqu Xiaoshi Oral Liquid for the Intestinal Microbiome of Children With Functional Dyspepsia
Brief Title: Influence of Shenqu Xiaoshi Oral Liquid on Intestinal Microbiome of Children With Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SQXS20220325
Record Dates: First submitted 2022-08-10; First posted 2022-08-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Dyspepsia; Child
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shenqu Xiaoshi Oral liquid (Experimental): Shenqu Xiaoshi Oral liquid will be taken orally.
  Interventions: Drug: Shenqu Xiaoshi Oral liquid

INTERVENTIONS:
Drug: Shenqu Xiaoshi Oral liquid — The dosage was determined by age: 3-4 years old, 5 ml/dose; 5-14 years old 10 ml/dose. Taken half an hour after meals, three times a day.
  Other Names: SXOL

SUMMARY:
It has been confirmed that treatment with Shenqu Xiaoshi Oral liquid (SXOL) effectively improves dyspeptic symptoms and is well tolerated. It is not inferior to domperidone syrup and leads to sustained improvement in Chinese children with functional dyspepsia (FD). This study aims to evaluate the possible regulatory effect of SXOL on intestinal microbiome in children with FD, further exploring its related mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients aged 3-14 years old;
2. Meeting ≥1 condition(s): (1)Postprandial fullness;(2)early satiation;(3)Epigastric pain or burning not associated with defecation;
3. Having symptoms at least 2 months and at least 4 days per month before diagnosis;
4. During the 2-wk lead-in period, no relevant drugs for the treatment of dyspepsia and anorexia were used, good eating habits have been established, and the FD symptoms still existed (symptom score≥3).
5. Informed consent was obtained from the parents/guardians of the participant. If the child was more than 8 years old, additional informed consent would be required from the participant.

Exclusion Criteria:

1. Anorexia and dyspepsia caused by certain drugs and confirmed organic diseases such as erosive gastritis, peptic ulcer, etc;
2. Severe malnutrition;
3. Serious primary diseases of the cardiovascular, nervous, respiratory, hepatobiliary and endocrine systems;
4. Mental disorders, intellectual disabilities, and/or communication impairments;
5. Lactose intolerant or allergic to the ingredients of Shenqu Xiaoshi Oral Liquid or Traditional Chinese medicine;
6. Probiotics or antibiotics within 4-wk;
7. Participated in a clinical trial within the past 12-wk;
8. Individuals deemed unsuitable for this clinical trial.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiome characteristics | Treatment for 2-week
  All subjects faeces will be collected and analyzed by high-throughput metagenomic sequencing to find the characteristics (e.g., the α and β diversity, the abundance of changed species) and composition of intestinal microbiome.
Intestinal microbiome metabolites | Treatment for 2-week
  Microbiome metabolites (e.g., short-chain fatty acid and bile acid) will be detected and analyzed by liquid chromatography-mass spectrometry (LC-MC) non-targeted metabolomics.
Levels of hormones | Treatment for 2-week
  e.g., Gastrin and Motilin
Levels of inflammatory cytokines | Treatment for 2-week
  e.g., TNF-α and IL-6
Clinical symptoms evaluation | Treatment for 1-week and 2-week
  Measured by a scale filling by subjects or their parents. The scale contains clinical symptoms of functional dyspepsia, such as postprandial fullness and early satiation. Scores range from 0 to 3 and higher scores represent more severe or more frequent.

CONTACTS AND LOCATIONS:
Overall Officials: Chundi Xu, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No